CLINICAL TRIAL: NCT06496217
Title: A Phase 1, Open-Label, Parallel-Group, Single Dose Adaptive Study to Evaluate the Safety and Pharmacokinetics of MBX 2109 in Adult Subjects With Normal and Impaired Renal Function
Brief Title: Safety and Pharmacokinetics Study of MBX 2109 in Adult Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: MBX-2H1003
Record Dates: First submitted 2024-06-12; First posted 2024-07-11 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single 900 µg dose of MBX 2109 (Experimental): A single, 900 µg dose of MBX 2109 will be administered subcutaneously in the abdomen
  Interventions: Drug: MBX 2109

INTERVENTIONS:
Drug: MBX 2109 — Group 1: Subjects with mild renal impairment (eGFR ≥ 60 and < 90 mL/min)
Drug: MBX 2109 — Group 2: Subjects with moderate renal impairment (eGFR ≥ 30 and < 60 mL/min)
Drug: MBX 2109 — Group 3: Subjects with severe renal impairment (eGFR < 30 mL/min), or kidney failure and not receiving dialysis
Drug: MBX 2109 — Group 4: Matched healthy subjects with normal renal function (eGFR ≥ 90 mL/min)

SUMMARY:
Evaluate the Safety and Pharmacokinetics of MBX 2109 in Adult Subjects with Normal and Impaired Renal Function

DETAILED DESCRIPTION:
A Phase 1, Open-Label, Parallel-Group, Single-Dose Adaptive Study to Evaluate the Safety and Pharmacokinetics of MBX 2109 in Adult Subjects with Normal and Impaired Renal Function

ELIGIBILITY:
Inclusion Criteria (all participants)

1. Willingness to adhere to the Protocol requirements as evidenced by a signed and dated informed consent form (ICF)
2. Subject is, as stated and in the opinion of the Investigator, willing and able to comply with the study drug regimen and all other study procedures and requirements, and is available for the duration of the study
3. Adult male or female, of at least 18 years of age, but not older than 80 years
4. Subject is willing to comply with the contraceptive requirements.
5. BMI ≥ 18.5 kg/m2 and < 40.0 kg/m2 at the time of Screening.
6. Light-, non- or ex-smoker
7. Has suitable venous access for blood sampling

   Subjects with Normal Renal Function (Group 4):
8. Medically healthy, in the opinion of an Investigator, with clinically insignificant Screening results (eg, laboratory profiles, medical history, vital signs, ECG, physical examination)
9. Normal renal function with eGFR ≥ 90 mL/min at Screening
10. Must match to the pooled mean age (± 10 years), BMI (within 20%) and gender (ratio should be similar) of mild, moderate, and severe (if applicable) renal impaired subjects at Screening.

    Subjects with Mild, Moderate, and Severe Renal Impaired Function (Groups 1, 2, and 3):
11. Considered clinically stable in the opinion of an Investigator
12. Presence of mild renal impairment (eGFR ≥ 60 and <90 mL/min), moderate renal impairment (eGFR ≥ 30 and <60 mL/min), or severe renal impairment (eGFR <30 mL/min) or kidney failure not receiving dialysis, at Screening: renal impairment should have been stable for at least 1 month prior to Screening.

Exclusion Criteria (All Participants)

1. Female who is lactating or breastfeeding
2. Female who is pregnant according to the pregnancy test at Screening or prior to study drug administration or planning to become pregnant before 90 days after the last study drug administration.
3. History of significant hypersensitivity to MBX 2109 or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
4. History of, or positive test for hepatitis B surface antigen (HbsAg), hepatitis C antibody (HCV Ab), or HIV antibody, at Screening.
5. Presence or history of any disorder that could interfere with completion of the study based on the opinion of an Investigator.
6. Intake of MBX 2109, or any investigational product (IP) in the 28 days prior to study drug administration.
7. Have urinary incontinence without catheterization
8. Receipt of blood products within 3 months prior to study drug administration.
9. Donation of 50 mL or more of blood in the 28 days prior to study drug administration
10. Donated 500 mL or more of blood within 56 days prior to study drug administration
11. Donated plasma within 2 weeks prior to Screening or donated platelets within 6 weeks prior to Screening.
12. Immunization with a Coronavirus Disease 2019 (COVID-19) vaccine in the 14 days prior to the first study drug administration.
13. Scheduled immunization with a COVID-19 vaccine during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason.
14. Use of St. John's wort in the 28 days prior to the first study drug administration.
15. Inclusion in a previous group for this clinical study
16. Any skin condition and/or tattoo that may interfere with the injection site evaluation.

    Subjects with Normal Renal Function (Group 4):
17. Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects.
18. History of significant gastrointestinal, liver, or kidney disease that may affect drug bioavailability.
19. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease.
20. Presence of clinically significant ECG abnormalities at the Screening visit, as defined by medical judgment.
21. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first study drug administration.
22. Supine or semi-supine blood pressure below 90/50 mmHg at the Screening visit
23. Supine or semi-supine blood pressure higher than 140/90 mmHg at the Screening visit (blood pressure readings greater than 140/90 mmHg may be retested if completed thought to be influenced by stress, at the discretion of the Investigator).
24. Supine or semi-supine pulse rate less than 40 beats per minute (bpm) or more than 100 bpm at Screening.
25. Any clinically significant illness in the 28 days before Day 1 of the study
26. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days before Day 1 of the study.
27. Use of over-the-counter (OTC) drugs and natural health products (eg, herbal remedies) at least 7 days (or 5-times the half-life of the drug, if longer) prior to study drug administration.
28. Use of any enzyme-modifying drugs, or drugs with effects on membrane transporters, including any strong cytochrome P450 3A4 and P-glycoprotein inducers and inhibitors in the previous 28 days before Day 1 of the study.

    Subjects with Mild, Moderate, and Severe Renal Impaired Function (Groups 1, 2, and 3):
29. History of renal transplant
30. Supine or semi-supine blood pressure below 90/50 mmHg at the Screening visit.
31. Supine or semi-supine blood pressure higher than 180/110 mmHg at the Screening visit.
32. Supine or semi-supine pulse rate less than 45 bpm or more than 110 bpm at Screening.
33. History or presence, in the opinion of an Investigator, of significant clinically unstable respiratory, cardiovascular, pulmonary, hepatic, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
34. Presence of poorly controlled Type 1 or Type 2 diabetes as defined by Hemoglobin A1c > 10%.
35. Presence of clinically significant physical examination, laboratory test, or ECG finding that, in the opinion of an Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results.
36. Subjects requiring treatment for renal impairment or other chronic disease (eg, well controlled diabetes, hypertension) must be on a stable treatment plan (medicines, doses, and regimens) for at least 14 days (except insulin) prior to study drug administration and during the entire study.
37. Positive Screening of alcohol and/or drugs of abuse at Screening or prior to study drug administration unless results can be explained by a prescription medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Maximum observed concentration (Cmax) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Area under the plasma concentration-time curve from time 0 to time of last quantifiable sample (AUC0-T) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Apparent clearance (CL/F) (MBX 2109 only) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Time to maximum concentration (Tmax) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Terminal elimination half-life (t1/2) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose
Apparent volume of distribution (Vz/F) (MBX 2109 only) | Baseline through Day 36
  Assess the plasma pharmacokinetics (PK) of MBX 2109 and MBX 2099 following a single 900 µg subcutaneous (SC) dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MBX Biosciences Investigational Site, Miami, Florida
  - MBX Bioscience Investigational Site, Tampa, Florida
  - MBX Biosciences Investigational Site, Minneapolis, Minnesota